CLINICAL TRIAL: NCT04959877
Title: Role of Health Education in the Semipresential Logopedic Treatment of the Patient With Oropharyngeal Dysphagia
Acronym: EDU-DIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-EDU-2021-50
Record Dates: First submitted 2021-06-20; First posted 2021-07-13 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed with oropharyngeal dysphagia who require speech therapy treatment for this reason and who have voluntarily opted for the blended treatment modality.
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: health education — data collect / Telemedicine

SUMMARY:
When reviewing the literature, the need to investigate the health education of patients with dysphagia and their family members / caregivers has been detected. Numerous articles mention or it can be inferred from them that an education or training has been carried out for the patient and caregivers, but the investigators have not found any that specifically focuses on this aspect of the intervention. Only in some Clinical Practice Guidelines is the need for health education included

ELIGIBILITY:
Inclusion Criteria:

* People between 18 and 99 years old diagnosed by videofluoroscopy of oropharyngeal dysphagia and who are candidates for speech therapy treatment for this reason.
* Knowledge of the language sufficient to understand the audiovisual material on health education available at: logopediasantpau.wordpress.com
* Have the necessary technological tools to carry out the telematic processing (electronic device with Internet access and WhatsApp) and know how to use them or have a family member / direct caregiver with basic technological skills.
* Signature of the informed consent

Exclusion Criteria:

* Moderate or severe cognitive impairment already known from the medical history or evaluated with the MoCA test in the absence of a family member or caregiver.
* Having undergone speech therapy treatment for oropharyngeal dysphagia in the last year.
* Not signing the informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with oropharyngeal dysphagia who require speech therapy
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Severity Rating Scale | up to 1 year
  Scale assessment by MBS ( 1 Non Oral - 7 Full oral intake)
Functional oral intake scale | up to 1 year
  Scale assessment (1nothing by mouth - 7 full oral intake)
Penetration Aspiration Scale | up to 1 year
  Scale Assessment by MBS (1 No airway penetration - 8 Airway aspiration, no cough)
Bolus Residual Scale | up to 1 year
  Scale Assessment by MBS (1 No residues - 6 Residue in Valleculae and posterior Pharyngeal wall and piriform sinus)

SECONDARY OUTCOMES:
SwalQOL | Up to 1 year
  Quality of life related to oropharyngeal dysphagia (11 Domains)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la santa creu i sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided